CLINICAL TRIAL: NCT05384548
Title: Can You Reduce Problematic Smartphone Use Through a Group Intervention: A Single Case Experimental Design
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We were unable to recruit and retain sufficient participants.
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020_Brett_Hayes_MRP
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Addiction, Smartphone
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Masking Description: Outcome measures will be collected electronically without involvement of the researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Problematic smart phone use course (Experimental)
  Interventions: Behavioral: Problematic smart phone use course

INTERVENTIONS:
Behavioral: Problematic smart phone use course — A 6 session, online, group-based, psychological course targetting problematic smart phone use.

SUMMARY:
This study will develop and conduct an initial, single-case, mixed-methods evaluation of a brief group intervention for mild and moderate problematic phone use.

ELIGIBILITY:
Inclusion Criteria:

-Self-identifies as struggling with problematic smart phone use

Exclusion Criteria:

* Actively experiencing suicidal or self-injurious thoughts, or have experienced these within the past year
* Already in a psychological therapy/intervention
* Planning a change of psychotropic medication during the research project.
* No access to video calling and/or slow internet connection speed
* A mental health condition that is not currently well managed/stable and therefore other interventions are likely to be more appropriate
* Does not own a smartphone that can record screen time
* Is not living in the UK, with access to services within the UK

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Change from pre-intervention (week 1) at post-intervention (week 10) on the Smartphone Addiction Scale -Short Version (SAS-SV). | Post-intervention (week 10)
  This measures smartphone addiction producing a score between 10 and 60, with higher scores indicating greater levels of addiction.

SECONDARY OUTCOMES:
Change from pre-intervention (week 1) at follow-up (week 18) on the Smartphone Addiction Scale -Short Version (SAS-SV). | Follow-up (week 18)
  This measures smartphone addiction producing a score between 10 and 60, with higher scores indicating greater levels of addiction.
Change from pre-intervention (week 1) at post-intervention (week 10) on the Depression, Anxiety and Stress Scale -21 item version (DASS-21). | Post-intervention (week 10)
  This measures levels of depression, anxiety and stress, producing a score between 0 for 42 each, with higher levels indicating greater severity.
Change from pre-intervention (week 1) at follow-up (week 18) on the Depression, Anxiety and Stress Scale -21 item version (DASS-21). | Follow-up (week 18)
  This measures levels of depression, anxiety and stress, producing a score between 0 for 42 each, with higher levels indicating greater severity.
Change from pre-intervention (week 1) at post-intervention (week 10) on the Multicultural Quality of Life Index. | Post-intervention (week 10)
  This measures of quality of life, producing a score between 1 and 10, with higher scores indicating greater quality of life.
Change from pre-intervention (week 1) at follow-up (week 18) on the Multicultural Quality of Life Index. | Follow-up (week 18)
  This measures of quality of life, producing a score between 1 and 10, with higher scores indicating greater quality of life.
Change in daily subjective units of distress from the baseline period (weeks 0 and 1) to the intervention period (weeks 2 to 9) | Intervention period (weeks 2 to 9)
  Single case analysis will compare daily subject units of distress ratings from the baseline period to the intervention period. Separate daily ratings, on a 0 to 100 scale, will be obtained for each of anxiety, stress, low mood, and tiredness, with higher ratings indicating higher levels.
Change in daily subjective units of distress from the baseline period (weeks 0 and 1) to the follow-up period (weeks 17 to 18) | Follow-up period (weeks 17 to 18)
  Single case analysis will compare daily subject units of distress ratings from the baseline period to the follow-up period. Separate daily ratings, on a 0 to 100 scale, will be obtained for each of anxiety, stress, low mood, and tiredness, with higher ratings indicating higher levels.
Change in daily phone use from the baseline period (weeks 0 and 1) to the intervention period (weeks 2 to 9) | Intervention period (weeks 2 to 9)
  Single case analysis will compare daily phone use from the baseline period to the intervention period. Daily use will be measured by screentime (in minutes) and number of pick-ups.
Change in daily phone use from the baseline period (weeks 0 and 1) to the follow-up period (weeks 17 to 18) | Follow-up period (weeks 17 to 18)
  Single case analysis will compare daily phone use from the baseline period to the follow-up period. Daily use will be measured by screentime (in minutes) and number of pick-ups.

OTHER OUTCOMES:
Qualitative interview | Week 18
  In week 18, a qualitative interview will be conducted, based on Elliot's Change Interview. This will explore participants' experiences of the intervention and perceptions of related change.

CONTACTS AND LOCATIONS:
Overall Officials: Brett Hayes, Principal Investigator — Canterbury Christ Church University; Fergal Jones, Study Director — Canterbury Christ Church University
Locations (1):
- Salomons Institute, Canterbury Christ Church University, Royal Tunbridge Wells, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No